CLINICAL TRIAL: NCT05890664
Title: Colchicine After Electrocardioversion for Atrial Fibrillation - The COLECTRO-AF Trial
Brief Title: Colchicine After Electrocardioversion for Atrial Fibrillation
Acronym: COLECTRO-AF
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss Heart Foundation (Other); Fondation Machaon, Switzerland, Genf (Unknown); Foundation for Cardiovascular Research Basel (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-00548, kt21sticherling
Record Dates: First submitted 2023-05-23; First posted 2023-06-06 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Atrial Fibrillation; Cardiac Arrhythmia
Keywords: Electrocardioversion; Colchicine
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double-blind, placebo-controlled trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A randomization list will be provided by the Clinical Trial Unit Basel to an unblinded person at the sponsor's site. The unblinded person will allocate the randomization numbers. Patients and research staff involved in patient recruitment, data management, outcome adjudication and data analyses will fully be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Study participants in the active study arm will receive a daily oral dose of 0.5 mg Colchicine for 3 months without a loading dose. The dose is recommended to be taken in the morning. There is no deviation from the usual treatment intake.
  Interventions: Drug: Colchicine
- Control Group (Placebo Comparator): Study participants in the placebo group will receive a matched placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine — Colchicine 0.5 mg (oral) once daily for 90 days. The chemical name for colchicine is (S)-N-(5,6,7,9-tetrahydro-1,2,3,10-tetramethoxy-9 oxobenzol[a]heptalen-7-yl) acetamide.
  Colchicine consists of pale yellow scales or powder. It is soluble in water, freely soluble in alcohol, and slightly soluble in ether.
  Arms: Experimental Group
Drug: Placebo — Matched placebo. Both the active drug and placebo will look similarly. The route and mode of administration is also similar to the active group.
  Arms: Control Group

SUMMARY:
The purpose of this study is to investigate whether a 3 month treatment course of low-dose Colchicine decreases the recurrence of Atrial fibrillation (AF) after electrocardioversion (ECV) in patients with AF.

DETAILED DESCRIPTION:
Atrial fibrillation is the most common cardiac arrhythmia worldwide and is associated with an increased risk of heart failure, stroke and death. Over the next 40 years the investigators expect another increase in the prevalence of atrial fibrillation with a risk of 1:3 in people over 65 years to develop atrial fibrillation. Electroconversion can occur in patients with atrial fibrillation reestablish sinus rhythm acutely with a controlled electrical shock. Unfortunately it is known however, that there is a short-term recurrence of atrial fibrillation in about 60%. This underlines that our current treatment options are inadequate. There is increasing evidence that inflammation is integral to initiation and maintenance of atrial fibrillation. Therefore, the researchers see inflammation as a possible therapeutic target to reduce the recurrence rate of atrial fibrillation after electroconversion. To test this hypothesis and to help patients, the investigators want to conduct the COLECTRO-AF study.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* ECG-documented AF prior to ECV
* Successful ECV with conversion of AF to sinus rhythm with persistent sinus rhythm ≥30 minutes after ECV
* Ability to give written informed consent

Exclusion Criteria:

* AF persistence after cardioversion or early AF recurrence within 30 minutes after ECV
* Any other rhythm than AF before cardioversion
* Pulmonary vein isolation within 3 months prior to ECV or pulmonary vein isolation planned within 3 months after ECV
* Known intolerance or hypersensitivity to Colchicine
* Any other absolute indication for Colchicine intake
* Intake of a strong inhibitor of CYP3A4 or P-Glycoprotein (clarithromycin, erythromycin, telithromycin, cyclosporine, ketoconazole or itraconazole)
* Serious gastrointestinal disease (severe gastritis or diarrhea)
* Clinically overt hepatic disease
* Severe renal disease (eGFR< 30ml/min/1.73m2)
* Clinically significant blood dyscrasia (e.g., myelodysplasia)
* Significant immunosuppression (e.g. due to transplantation or rheumatic disease)
* Pregnant or breastfeeding women, or women of child-bearing potential who do not use a highly effective form of birth control
* Life expectancy <1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Estimated)
Dates: Start 2024-04-14 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Number of atrial fibrillation (AF) recurrence | within 6 month after electrocardioversion
  The primary outcome of AF recurrence within 6 months will be assessed based on the ECG (electrocardiogram) documentation of any AF. If a patient reports symptoms of AF recurrence in between the study visits, the research staff will obtain an ECG documentation. The outcome will only be valid if AF recurrence is documented by an ECG.

SECONDARY OUTCOMES:
Number of atrial fibrillation (AF) recurrence | within 1 month after electrocardioversion
  The secondary outcome of AF recurrence within 1 months will be assessed based on the ECG (electrocardiogram) documentation of any AF. If a patient reports symptoms of AF recurrence in between the study visits, the research staff will obtain an ECG documentation. The outcome will only be valid if AF recurrence is documented by an ECG.
Number of atrial fibrillation (AF) recurrence | within 3 month after electrocardioversion
  The secondary outcome of AF recurrence within 3 months will be assessed based on the ECG (electrocardiogram) documentation of any AF. If a patient reports symptoms of AF recurrence in between the study visits, the research staff will obtain an ECG documentation. The outcome will only be valid if AF recurrence is documented by an ECG.
Time to first redo electrocardioversion | up to 6 month
  Time to first redo electrocardioversion
Use of antiarrhythmic drugs | within 6 month after electrocardioversion
  Assessment of medication intake by study staff Vaughan-Williams classification class 1 and 3 of antiarrhythmic drugs will be documented (1 = sodium channel blockade, 3 = potassium channel blockade)
Number of survived participants without an unplanned hospital stay | up to 6 month
  Number of survived participants without an unplanned hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Krisai, PD Dr. med., Principal Investigator — University Hospital, Basel, Switzerland
Locations (8):
- Switzerland (8):
  - Cantonal Hospital Baselland (KSBL), Bruderholz, Basel-Landschaft
  - University Hospital Basel, Basel
  - University Hospital Bern, Bern
  - Lausanne University Hospital, Lausanne
  - Lucerne Cantonal Hospital, Lucerne
  - Cantonal Hospital Olten, Olten
  - Herzpraxis am Rhein, Rheinfelden
  - Solothurner Spitäler AG, Solothurn